CLINICAL TRIAL: NCT00122135
Title: A Culturally Sensitive Values-Guided Aid for End of Life Decision-Making
Acronym: Aim3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 02-224
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Congestive Heart Failure; Chronic Obstructive Pulmonary Disease; Cirrhosis; Colon Carcinoma; Lung Cancer; Chronic Kidney Disease
Keywords: end-of-life care; clinical decision-making; values inventory; racial disparities
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Fibrosis; Colonic Neoplasms; Lung Neoplasms; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients without Values Inventory (VI) (No Intervention): Clinic encounter w/physician & patient and/or surrogate - Patients who did not receive the VI prior to their physician clinic encounter
- Patients with Values Inventory (VI) (Experimental): Clinic encounter w/physician & patient and/or surrogate - Patients who completed the VI prior to their physician clinic encounter
  Interventions: Other: Values Inventory (VI)

INTERVENTIONS:
Other: Values Inventory (VI) — The Values Inventory was given to patients for self-administration while they were awaiting their clinic appointment. They were instructed to bring it to their physician's attention right at the beginning of their clinic visit.
  Arms: Patients with Values Inventory (VI)

SUMMARY:
The goal of this research agenda is to improve the quality of end-of-life care by explicitly identifying values that will guide the decision-making process, with a particular emphasis on the role of ethnic, racial and cultural factors.

DETAILED DESCRIPTION:
Background: End-of-life decision-making is an important aspect of providing quality healthcare, especially for the elderly population. Increasingly, the appropriateness of many of these decisions is being questioned. Some invasive procedures done in seriously ill patients do not significantly alter their course, many patients die without having pain or other symptoms addressed, and families may feel dissatisfied with the care provided. Additionally, there are striking racial/ethnic disparities in end-of-life care.

Objectives: The explicit identification of values that guide medical decision-making could improve the decision-making process for end-of-life care for patients of all races/ethnicities. 1) We will directly compare, critically assess, and revise two Values Histories on the basis of qualitative data derived from individual interviews with racially/ethnically diverse patients and surrogates, and explore patients', surrogates', and physicians' values, preferences and concerns that guide decision-making about medical interventions at the end-of-life. 2) We will then adapt the existing Values Histories into a clinically practical tool, the Values Inventory discussion aid. 3) We will conduct preliminary testing of this tool to be used in physician-patient or physician-surrogate encounters to improve and facilitate decisions about end-of-life care.

Methods: To complete Objective 3 we will conduct a pilot randomized trial of the developed Values Inventory discussion aid to test the feasibility of using it in clinical practice. This clinicaltrials.gov number applies to Objective 3 of IIR-02-224 only (as the complete study is a mixed-methods study with several different arms and enrollment goals). Eligible patients are at risk for 6-12-month mortality with one of the following diagnoses: congestive heart failure, with ejection fraction of less than 25%; severe chronic obstructive pulmonary disease/emphysema with dependence on oxygen; chronic liver disease with cirrhosis and ascites; colon carcinoma with liver metastases; or non-small cell cancer of the lung, stage III or IV, and patients with chronic kidney disease on renal replacement therapy, with previous hospitalization. All (patient) participants are age 55 years or older and are recruited through the clinics/wards at the Houston VAMC. Surrogates are surrogates of patients with such conditions; physicians are generalists and medical subspecialists. All participants are African American, Hispanic, or White, reflecting the 3 major races/ethnicities at the Houston VAMC.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be at risk for 6-12 month mortality and have one of the following diagnoses:

  * congestive heart failure, with ejection fraction of <25%;
  * severe chronic obstructive pulmonary disease/emphysema with dependence on oxygen;
  * chronic liver disease with cirrhosis and ascites;
  * colon carcinoma with liver metastases; or
  * non-small cell cancer of the lung, stage III or IV
  * chronic kidney disease on renal replacement therapy, with previous hospitalization
* All participants will be age 55 years or older and will be recruited through the clinics at the Houston VAMC.

Exclusion Criteria:

* Patients with dementia
* Patients less than 55 years old

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula K. Braun, MD MPH, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E DeBakey VA Medical Center, Houston, Texas, United States

REFERENCES:
- [Result] Braun UK, Beyth RJ, Ford ME, McCullough LB. Defining limits in care of terminally ill patients. BMJ. 2007 Feb 3;334(7587):239-41. doi: 10.1136/bmj.39048.475046.68. PMID 17272566
- [Result] Braun UK, Beyth RJ, Ford ME, McCullough LB. Voices of African American, Caucasian, and Hispanic surrogates on the burdens of end-of-life decision making. J Gen Intern Med. 2008 Mar;23(3):267-74. doi: 10.1007/s11606-007-0487-7. Epub 2008 Jan 3. PMID 18172738
- [Result] Braun UK, Kunik ME, Pham C. Treating depression in terminally ill patients can optimize their physical comfort at the end of life and provide them the opportunity to confront and prepare for death. Geriatrics. 2008 Jun;63(6):25-7. PMID 18512998
- [Result] Braun UK, McCullough LB, Beyth RJ, Wray NP, Kunik ME, Morgan RO. Racial and ethnic differences in the treatment of seriously ill patients: a comparison of African-American, Caucasian and Hispanic veterans. J Natl Med Assoc. 2008 Sep;100(9):1041-51. doi: 10.1016/s0027-9684(15)31442-5. PMID 18807433
- [Result] Braun UK, Naik AD, McCullough LB. Reconceptualizing the experience of surrogate decision making: reports vs genuine decisions. Ann Fam Med. 2009 May-Jun;7(3):249-53. doi: 10.1370/afm.963. PMID 19433843
- [Result] Braun UK, Ford ME, Beyth RJ, McCullough LB. The physician's professional role in end-of-life decision-making: voices of racially and ethnically diverse physicians. Patient Educ Couns. 2010 Jul;80(1):3-9. doi: 10.1016/j.pec.2009.10.018. Epub 2009 Nov 30. PMID 19948388
- [Result] Braun UK, Ford ME, McCullough L, Beyth RJ. Discussing End-of-Life Decision Making: Views of Racially and Ethnically Diverse Physicians. [Abstract]. The Journal of Nutrition, Health & Aging. 2006 Aug 1; 10(4):332.
- [Result] Nambiar A, McCullough L, Ford M, Beyth R, Braun UK. Discussing End-of-Life Decision Making: Views of Racially and Ethnically Diverse Physicians. [Abstract]. The Gerontologist. 2006 Oct 1; 46(Special Issue 1):402.
- [Result] Braun U, Morgan RO, Ford ME, Beyth RJ. Who gets what? Race/ethnicity matter for treatment of seriously ill veterans. [Abstract]. Journal of the American Geriatrics Society. 2006 Apr 1; 54(S4):S180.
- [Result] Braun U, McCullough L, Ford M, Espadas D, Beyth R. End-of-life care across race and ethnicities: Voices of patients, surrogates, and physicians. [Abstract]. Journal of the American Geriatrics Society. 2005 Apr 1; 53(s1):S137-8.
- [Result] Pham C, Braun UK. Racial and Ethnic Differences in End-of-Life Care for Patients with End-Stage Renal Disease. [Abstract]. Journal of pain and symptom management. 2009 Mar 1; 37(3):556-557.
- [Result] Braun UK, Beyth RJ, Ford ME, Espadas D, McCullough LB. Decision-making styles of seriously ill male Veterans for end-of-life care: Autonomists, Altruists, Authorizers, Absolute Trusters, and Avoiders. Patient Educ Couns. 2014 Mar;94(3):334-41. doi: 10.1016/j.pec.2013.10.013. Epub 2013 Nov 19. PMID 24365071
- [Result] Braun UK, McCullough LB. Preventing life-sustaining treatment by default. Ann Fam Med. 2011 May-Jun;9(3):250-6. doi: 10.1370/afm.1227. PMID 21555753
- [Result] Menon S, McCullough LB, Beyth RJ, Ford ME, Espadas D, Braun UK. Feasibility of Using a Values Inventory as a Discussion Aid about End-of-Life Care. Poster session presented at: Gerontological Society of America Annual Scientific Meeting; 2010 Nov 21; New Orleans, LA.
- [Result] Menon S, McCullough LB, Beyth RJ, Ford ME, Espadas D, Braun UK. Use of a values inventory as a discussion aid about end-of-life care: A pilot randomized controlled trial. Palliat Support Care. 2016 Aug;14(4):330-40. doi: 10.1017/S1478951515001091. Epub 2015 Oct 13. PMID 26458331

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With VI: patients / surrogates who did receive the Values Inventory prior to their clinic appointment
  Values history discussion w/physician & patient/surrogate: 128 patient/physician values history discussions were taped, also 4 case studies with surrogates were completed.
- Patients Without VI: Patients who did not receive the Values Inventory prior to their clinic visit
Period: Overall Study
Arm/Group | Patients With VI | Patients Without VI
Started | 60 | 60
Completed | 57 | 60
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With VI: Patients who filled out the Values History prior to their clinic appointment
- Patients Without VI: Patients who did not receive the Values History prior to their clinic appointment (usual care)
- Total: Total of all reporting groups
Arm/Group | Patients With VI | Patients Without VI | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 27 | 57
  >=65 years | 30 | 33 | 63
Age, Continuous [Mean (Full Range); unit: years] | 66.4 [55 to 85] | 68.4 [56 to 84] | 67.4 [55 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 60 | 60 | 120
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Presence of Discussions About End of Life Care Goals/Wishes
Description: Qualitative content analysis of physician-patient encounters regarding presence of any type of discussion about end of life care goals/wishes
Time Frame: immediate
Measure: Number; unit: participants
Arm/Group | Patients With VI | Patients Without VI
Number analyzed (Participants) | 57 | 60
participants | 13 | 8
Statistical Analysis 1: Comparison: Patients With VI vs Patients Without VI; Test type: Superiority or Other; p = .77, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: There was only a one-time physician-patient encounter for this minimum risk study and any adverse event would have been reported immediately on the day of the encounter. There was no systematic assessment for AE.
Description: No patient reported an adverse event at the time of the study (immediately before/after physician - patient encounter. Nobody reported any adverse events later to study personnel.
Groups:
- Patients With VI: Clinic encounter w/physician & patient and/or surrogate - Patients who completed the VI prior to their physician clinic encounter
  Clinic encounter w/physician & patient and/or surrogate: 128 patient/physician values history discussions were taped, also 4 case studies with surrogates were completed.
- Patients Without VI: Clinic encounter w/physician & patient and/or surrogate - Patients who did not receive the VI prior to their physician clinic encounter
  Clinic encounter w/physician & patient and/or surrogate: 128 patient/physician values history discussions were taped, also 4 case studies with surrogates were completed.
Arm/Group | Patients With VI | Patients Without VI
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
Difficulties in recruiting enough surrogates led to abandoning having a surrogate arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes